CLINICAL TRIAL: NCT06835920
Title: Alcohol Labeling Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-1218b; R01AA030548 (NIH)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Front-of-package health warning (Experimental)
  Interventions: Behavioral: Front-of-package health warning
- Control label (Other)
  Interventions: Behavioral: Control label

INTERVENTIONS:
Behavioral: Front-of-package health warning — Participants will receive 3 different health warnings about alcohol consumption. The warnings will discuss health risks of alcohol including cancer, high blood pressure, and scarring of the liver. Labels will be placed on the front of participants' alcohol containers.
  Arms: Front-of-package health warning
Behavioral: Control label — Participants will receive a label displaying a barcode. Labels will be placed on the front of participants' alcohol containers.
  Arms: Control label

SUMMARY:
This study aims to examine the effects of new front-of-package alcohol warnings on alcohol consumption. Participants will be randomly assigned to either new front-of-package health warnings or control labels. Participants will bring in their own alcohol to weekly study visits and take home the alcohol to consume as usual. Participants will receive study labels on their alcohol containers per their assigned trial arm.

DETAILED DESCRIPTION:
This study aims to determine whether new front-of-package health warnings on alcohol containers lead to less alcohol consumption and improve consumer understanding about the harms of alcohol. We aim to enroll approximately 720 adults ages 21 years and older who report consuming alcohol at least once per week.

After providing informed consent, participants will be randomly assigned to receive new front-of-package health warnings or control labels.

Participants will attend 3 in-person study visits spaced approximately 1 week apart. Participants in the warnings arm will receive a health warning applied to the front of their alcohol containers at each of the weekly visits for a total of 3 unique warnings during the study. Warnings will be applied in counterbalanced order. Participants in the control arm will receive one label during the study.

Participants will report the number of drinks they consumed daily via text message and will complete 4 computer surveys spaced approximately 1 week apart.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 21 years and older
* Not identified as having possible alcohol dependence
* Consumed alcohol at least once per week during the past 4 weeks
* At least half of alcohol consumed each week is from store-bought containers
* Willing to bring 8 days' worth of alcohol to 3 in-person study visits
* Not pregnant, breastfeeding, or trying to get pregnant
* Able to take surveys in English
* Willing to respond to text messages daily for 3 weeks
* Not living in the same household as anyone else in the study

Exclusion Criteria:

- Not living in US

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of alcoholic drinks consumed | Assessed daily for 21 days, starting the day after enrollment.
  Measured using the following item "How many drinks did you have yesterday? If you're not sure, make your best guess. By 'yesterday,' we mean before you went to bed, even if the drinking happened after midnight. One drink is equivalent to a 12-ounce beer, a 5-ounce glass of wine, or a drink with one shot of liquor." Participants will respond with the number of drinks they consumed.

SECONDARY OUTCOMES:
Intentions to limit drinking | Assessed 4 times approximately 1-week apart, starting on the day of enrollment.
  Measured using 3 survey items: 1) "How interested are you in drinking no more than x drinks in the next week?" 2) "How much do you plan to have no more than x drinks in the next week?" and 3) "How likely are you to have no more than x drinks in the next week?" where x = 7 if the participant's sex at birth is female, 14 otherwise. Response options are on a 5-point scale with lowest endorsement coded as 1 and highest endorsement coded as 5. Researchers will average responses to the 3 items. Higher scores indicate greater intentions to limit drinking.
Forgoing a drink | Assessed approximately 1 week, 2 weeks, and 3 weeks after enrollment.
  Measured using 5 survey items asking participants how often they chose to forgo a drink during the study (e.g., "In the last 7 days, how often have you stopped yourself from having an alcoholic drink because you wanted to cut back?"). Response options are on a 5-point scale ranging from "Never" coded as 0, to "10 or more times", coded as 10. Researchers will average responses to the 5 items. Higher scores indicate greater frequency of forgoing a drink.
Maximum number of drinks in a day | Assessed daily for 21 days, starting the day after enrollment.
  Participants will report the number of drinks they had yesterday using the following item "How many drinks did you have yesterday?" For each participant, researchers will calculate the maximum number of drinks in a day as the highest number of drinks participants report consuming in one day during the study period.
Proportion of days drinking | Assessed daily for 21 days, starting the day after enrollment.
  Participants will report the number of drinks they had yesterday using the following item "How many drinks did you have yesterday?" The proportion of days drinking will be calculated as the number of days participants report consuming alcohol during the study divided by the total number of days they report their alcohol consumption during the study. Missing data will be excluded from both the numerator and denominator.
Perceived control over drinking | Assessed approximately 1 week, 2 weeks, and 3 weeks after enrollment.
  Measured using 1 survey item: "Did the labels make you feel...?" where response options are "Less in control of your drinking" "Neither less nor more in control of your drinking" and "More in control of your drinking." Responses will be coded as increasing control (1) vs. reducing control or neither increasing nor reducing (0).
Learning something new | Assessed once, approximately 21 days after enrollment.
  Measured using 1 survey item: "Did you learn something new from the labels?" where response options are "Yes" (coded as 1) and "No" (coded as 0).
Knowledge of harms from alcohol in warnings | Assessed once, approximately 21 days after enrollment.
  Measured using 3 survey items: "How does having 2 alcoholic drinks a day affect the risk of [cancer/ scarring of the liver/ high blood pressure]?" Response options include "Decreases risk" "No effect" "Increases risk" and "Not sure." Knowledge will be coded as correct if participants select "Increases risk" and incorrect if participants select any other option. Participants will receive a correct overall knowledge score only if they answer all 3 items correctly.
Reminding of harms of alcohol | Assessed 4 times approximately 1-week apart, starting on the day of enrollment.
  Measured using 1 survey item: "How much did the labels remind you that drinking alcohol can be harmful?" Response options are on a 5-point scale ranging from "Not at all", coded as 1 to "A great deal", coded as 5. Higher scores indicate greater reminding of harms of alcohol.
Perceived likelihood of harms from alcohol | Assessed 4 times approximately 1-week apart, starting on the day of enrollment.
  Measured using the item: "What is the chance that drinking 2 [standard drinks of alcohol type] a day will cause you to have health problems one day?" Participants will answer the question 4 times, once about 4 types of alcohol: beer, wine, hard seltzer, and liquor. Response options are on a 5-point scale ranging from "No chance", coded as 1 to "High chance", coded as 5. Responses to the 4 questions will be averaged. Higher scores indicate greater perceived likelihood of having health problems caused by alcohol.
Perceived healthfulness of alcohol | Assessed 4 times approximately 1-week apart, starting on the day of enrollment.
  Measured using the item: "How healthy or unhealthy is [alcohol type]?" Participants will answer the question 4 times, once about 4 types of alcohol: beer, wine, hard seltzer, and liquor. Response options are on a 5-point scale ranging from "Very unhealthy", coded as 1 to "Very healthy", coded as 5. Responses to the 4 questions will be averaged. Higher scores indicate greater perceived healthfulness of alcohol.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC study office, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT06835920/Prot_SAP_001.pdf